CLINICAL TRIAL: NCT02474355
Title: Open Label, Multinational, Multicenter, Real World Treatment Study of Single Agent AZD9291 for Patients With Advanced/Metastatic Epidermal Growth Factor Receptor (EGFR) T790M Mutation-Positive Non-Small Cell Lung Cancer (NSCLC) Who Have Received Prior Therapy With an EGFR Tyrosine Kinase Inhibitor (EGFR-TKI)
Brief Title: Real World Treatment Study of AZD9291 for Advanced/Metastatic EGFR T790M Mutation NSCLC
Acronym: ASTRIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5160C00022
Record Dates: First submitted 2015-05-27; First posted 2015-06-17 (Estimated); Results first posted 2021-10-25 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer
Keywords: NSCLC; EGFRm; T790M
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD9291 (Experimental): Single arm of AZD9291, starting dose of 80mg
  Interventions: Procedure: T790M+ Testing; Procedure: Baseline Visit Blood & Urine Testing; Procedure: Baseline ECG; Procedure: Visual Slit-Lamp Testing; Drug: AZD9291 Dosing

INTERVENTIONS:
Procedure: T790M+ Testing — If a previous lab report is unavailable, the patient will need to have T790M+ testing.
Procedure: Baseline Visit Blood & Urine Testing — Blood count and standard chemistry testing to ensure patient meets inclusion/exclusion criteria
Procedure: Baseline ECG — ECG to ensure absence of any cardiac abnormality
Procedure: Visual Slit-Lamp Testing — Slit-lamp testing performed to ensure patients do not have any eye abnormalities or symptoms
Drug: AZD9291 Dosing — Patients to be provided with AZD9291 every 6 weeks (+/- 7 days)

SUMMARY:
The aim of this study is to assess the efficacy and safety of single agent AZD9291 in a real world setting in adult patients with advanced or metastatic, epidermal growth factor receptor (EGFR) T790M mutation-positive Non-Small Cell Lung Cancer (NSCLC), who have received prior EGFR-tyrosine kinase inhibitor (TKI) therapy.

DETAILED DESCRIPTION:
Objective: The primary objective of this study is to assess the efficacy and safety of single agent AZD9291 in a real world setting in adult patients with advanced or metastatic, epidermal growth factor receptor (EGFR) T790M mutation-positive Non-Small Cell Lung Cancer (NSCLC), who have received prior EGFR-tyrosine kinase inhibitor (TKI) therapy.

Study site(s) and number of patients planned: Approximately 1500 patients will be recruited in Europe. The recruitment will be increased beyond that as the study will expand in other regions of the world (America, Asia).

Study Design This will be an open-label, single-arm, multinational, multicenter, real world treatment study.

Target patient population: Adult patients (fulfilling the definition of "age of majority" per local regulations) with locally advanced (stage IIIB) or metastatic (stage IV) NSCLC with confirmed T790M mutation, who have received prior EGFR-TKI therapy.

Investigational product (IP), dosage, and mode of administration: AZD9291 is an oral, potent, selective, irreversible inhibitor of both EGFR-TKI sensitising and resistance mutations in NSCLC with a significant selectivity margin over wild-type EGFR. AZD9291 will be administered orally as one 80 mg tablet once a day.

Duration of IP administration: Patients may continue to receive AZD9291 as long as they continue to show clinical benefit, as judged by the investigator, and in the absence of discontinuation criteria). The study will be closed in each participating country as soon as possible following national reimbursement of AZD9291 in that country (up to a max of 90 days post reimbursement). Enrolment will be closed within 6 months after market license approval in that country or at national reimbursement, whichever is sooner. Patients withdrawing from the treatment prior to national reimbursement will be followed up as part of this study. Patients on treatment will receive commercial supply until documented disease progression as per investigator assessment.

In the event that national reimbursement should not be granted following a reasonable time after market license approval in the country, the study will be closed in a maximum period of 18 months after the last patient is enrolled in that country. If applicable, timelines for conversion to commercial drug will be agreed with local bodies which may include regulatory agencies, ethics committees, and institutions. Patient will be followed until death or lost to follow-up.

Study measures: Data collected will include patient demographics, information needed to determine patient eligibility (including medical history, past and current disease characteristics, and tumor EGFR mutational status), AZD9291 exposure, investigator-reported efficacy (including tumor response and disease progression), overall survival (OS), and safety (including serious adverse events [SAEs], adverse events leading to dose modification, and adverse events of special interest [interstitial lung disease/pneumonitis-like events, and QTc prolongation events]).

Statistical methods: All data will be presented for the overall full analysis/evaluable set, and also by cohorts defined by number and type of previous treatment lines for the advanced disease. Descriptive statistics will be used for all variables, as appropriate. Continuous variables will be summarised by the number of observations, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarised by frequency counts and percentages for each category. OS and PFS will be summarized using Kaplan-Meier estimates of the median time to death or censoring and quartiles together with their 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent by the patient or legally acceptable representative prior to any study-specific procedures
2. Adults (according to each country regulations for age of majority)
3. Locally advanced (stage IIIB) or metastatic (stage IV) EGFRm NSCLC, not amenable to curative surgery or radiotherapy, with confirmation of the presence of the T790M mutation
4. Prior therapy with an EGFR-TKI. Patients may have also received additional lines of treatment
5. World Health Organization (WHO) performance status 0-2
6. Adequate bone marrow reserve and organ function as demonstrated by complete blood count, biochemistry in blood and urine at baseline (please refer to IB for guidance)
7. ECG recording at baseline showing absence of any cardiac abnormality as per exclusion criterion #6
8. Female patients of childbearing potential must be using adequate contraceptive measures, must not be breast feeding, and must have a negative pregnancy test prior to start of dosing. Otherwise, they must have evidence of nonchildbearing potential
9. Male patients must be willing to use barrier contraception, i.e., condoms

Exclusion Criteria:

1. Previous (within 6 months) or current treatment with AZD9291
2. Patients currently receiving (or unable to stop use at least 1 week prior to receiving the first dose of AZD9291) any treatment known to be potent inhibitors or inducers of cytochrome P450 (CYP) 3A4
3. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, active infection including hepatitis B, hepatitis C, and human immunodeficiency virus, or significantly impaired bone marrow reserve or organ function, including hepatic and renal impairment, which in the investigator's opinion would significantly alter the risk/benefit balance.
4. Patient with symptomatic central nervous system (CNS) metastases who is neurologically unstable or has required increasing doses of steroids to manage CNS symptoms within the 2 weeks prior to start AZD9291 administration;
5. Past medical history of ILD, drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD
6. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTcF) > 470 ms using Fredericia's formula :
   2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block)
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events
7. Any unresolved toxicity from prior therapy CTCAE > grade 3 at the time of starting treatment
8. History of hypersensitivity to excipients of AZD9291 or to drugs with a similar chemical structure or class to AZD9291

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3017 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (137):
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, CABA
- Australia (5):
  - Research Site, Bedford Park
  - Research Site, East Melbourne
  - Research Site, Kurralta Park
  - Research Site, Randwick
  - Research Site, Waratah
- Austria (4):
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Leuven
- Brazil (9):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Florianópolis
  - Research Site, Ijuí
  - Research Site, Itajaí
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo
- Canada (10):
  - Research Site, Calgary, Alberta
  - Research Site, Burnaby, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Regina, Saskatchewan
- China (34):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Nantong
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiahzhuang
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Yancheng
  - Research Site, Yangzhou
  - Research Site, Yantai
  - Research Site, Zhengzhou
- Research Site, Vejle, Denmark
- Research Site, Dublin, Ireland
- Italy (22):
  - Research Site, Ancona
  - Research Site, Avellino
  - Research Site, Bari
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Cagliari
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Lecce
  - Research Site, Livorno
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Palermo
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Udine
  - Research Site, Verona
- Saudi Arabia (2):
  - Research Site, Dammam
  - Research Site, Riyadh
- South Korea (16):
  - Research Site, Anyang
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gangneung-si
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, Jeonnam
  - Research Site, JinJoo
  - Research Site, Seogu
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Ulsan
- Spain (16):
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Castellon
  - Research Site, Donostia / San Sebastian
  - Research Site, Jaén
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, León
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza
- Sweden (2):
  - Research Site, Örebro
  - Research Site, Uppsala
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (5):
  - Research Site, Antrim
  - Research Site, London
  - Research Site, Norwich
  - Research Site, Poole
  - Research Site, Wolverhampton

REFERENCES:
- [Derived] Zhou Q, Zhang HL, Jiang LY, Shi YK, Chen Y, Yu JM, Zhou CC, He Y, Hu YP, Liang ZA, Pan YY, Zhuo WL, Song Y, Wu G, Chen GY, Lu Y, Zhang CY, Zhang YP, Cheng Y, Lu S, Wang CL, Zhou JY, Liu YP, He JX, Wang J, Wu YL. Real-world evidence of osimertinib in Chinese patients with EGFR T790M-positive non-small cell lung cancer: a subgroup analysis from ASTRIS study. J Cancer Res Clin Oncol. 2023 Sep;149(12):10771-10780. doi: 10.1007/s00432-023-04923-8. Epub 2023 Jun 14. PMID 37316692
- [Derived] Cheema P, Cho BC, Freitas H, Provencio M, Chen YM, Kim SW, Wu YL, Passaro A, Martin C, Tiseo M, Chang GC, Park K, Solomon B, Burghuber O, Laskin J, Wang Z, Lee SY, Hu Y, Vansteenkiste J, Zhang HL, Hanrahan E, Geldart T, Taylor R, Servidio L, Li J, Marinis F. A real-world study of second or later-line osimertinib in patients with EGFR T790M-positive NSCLC: the final ASTRIS data. Future Oncol. 2023 Jan;19(1):61-75. doi: 10.2217/fon-2022-0919. Epub 2023 Jan 19. PMID 36656302
- [Derived] Leighl NB, Kamel-Reid S, Cheema PK, Laskin J, Karsan A, Zhang T, Stockley T, Barnes TA, Tudor RA, Liu G, Owen S, Rothenstein J, Burkes RL, Iqbal M, Spatz A, van Kempen LC, Izevbaye I, Laurence D, Le LW, Tsao MS. Multicenter Validation Study to Implement Plasma Epidermal Growth Factor Receptor T790M Testing in Clinical Laboratories. JCO Precis Oncol. 2020 Nov;4:520-533. doi: 10.1200/PO.19.00335. PMID 35050743
- See also: D5160C00022 Clinical Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00022&attachmentIdentifier=dd920aaa-edfe-410c-9fae-e649b1f11351&fileName=223048_D5160C00022_CSP_Final_(deidentified).pdf&versionIdentifier=
- See also: D5160C00022 Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00022&attachmentIdentifier=e2241d73-0d0f-4439-b968-f6ed09f8d283&fileName=223048_D5160C00022_SAP_and_Addendum_Final_(deidentified).pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met all the inclusion and none of the exclusion criteria received treatment in a total of 209 centres in 16 countries. The study started on 18 September 2015 and primary completion date was 18 April 2019.
Pre-assignment Details: During the screening period (28 days), eligible participants signed the informed consent. All the study assessments were performed as per the schedule of assessment. Out of 3017 patients enrolled with treatment dose assigned, 3 died (due to disease progression) prior to starting treatment.
Groups:
- Osimertinib: All participants received oral 80 mg tablet once a day (the dose could be reduced to 40 mg for management of osimertinib-related toxicities)
Period: Overall Study
Arm/Group | Osimertinib
Started | 3014
Completed (Participants who withdrew from the study owing to study closure in their country. The participants received the study drug at time of study closure and continued treatment with reimbursed commercial drug or in a local patient support program, those who had discontinued study drug at study closure had their survival follow-up stopped.) | 1386
Not Completed | 1628
Not completed — Other | 43
Not completed — Eligibility Criteria not Fulfilled | 2
Not completed — Lost to Follow-up | 98
Not completed — Withdrawal by Subject | 124
Not completed — Death | 1361

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who received at least one dose of study treatment.
Arm/Group | Osimertinib
Number analyzed (Participants) | 3014
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1798
  >=65 years | 1216
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1927
  Male | 1087
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2085
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 897
  More than one race | 0
  Unknown or Not Reported | 11
Country [Count of Participants; unit: Participants]
  Argentina | 30
  Australia | 31
  Austria | 46
  Belgium | 31
  Brazil | 88
  Canada | 99
  China | 1350
  Denmark | 6
  Ireland | 10
  Italy | 510
  Saudi Arabia | 3
  South Korea | 466
  Spain | 131
  Sweden | 7
  Taiwan | 188
  United Kingdom | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time, in months from the date of first dose of Osimertinib until death due to any cause, or at last documented contact with participant status "alive" (in this study any participants alive at study discontinuation, or lost to follow-up was considered being censored at study discontinuation date or at the last known date participant was alive). OS was summarized using a Kaplan-Meier (KM) estimate of the median time to death or censoring together with their 95% confidence intervals.
Time Frame: From the date of first dose of Osimertinib until the date of death (due to any cause) or last participant contact [up to 43 months]
Population: The full analysis set included all participants who received at least one dose of study treatment. No statistical tests were performed, the statistical analyses were descriptive.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib
Number analyzed (Participants) | 3014
Months | 22.8 [21.6 to 23.8]

2. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Safety assessment of Osimertinib was analyzed by evaluating AEs and SAEs.
Time Frame: From screening to progression follow-up [every 6 weeks +/- 1 week] relative to the date of enrolment until the end of study [up to 43 months]
Population: The full analysis set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 3014
Participants
  AE of special interest (AESI) or SAE | 923
  AESI or SAE a causally related to Osimertinib | 338
  AE leading to dose modification | 414
  AE leading to discontinuation | 191
  AESI | 113
  AESI causally related to Osimertinib | 89
  SAE | 657
  SAE causally related to Osimertinib | 95
  AE leading to death | 152
  AE leading to death causally related to Osimertinib | 19

3. Secondary Outcome: Progression Free Survival
Description: PFS was defined as the time, in months from first dose of AZD9291/ost/study drug/ study treatment until the date of disease progression or death in the absence of progression. Participants who had not progressed or died at study discontinuation were censored at the time of the latest date of disease assessment. PFS was summarized using KM estimates of the median time to progression or death with their 95% confidence intervals.
Time Frame: From the date of first dose of Osimertinib until disease progression or death in the absence of progression [up to 43 months]
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib
Number analyzed (Participants) | 3014
Months | 11.1 [11.0 to 12.0]

4. Secondary Outcome: Time to Treatment Discontinuation (TTD)
Description: TTD or death was assessed as a supportive summary to PFS and defined as the time from the date of the first dose of osimertinib in the study until the date of osimertinib discontinuation or death, regardless of the reason for discontinuation. TTD was summarized using KM estimates of the median times to progression or death or treatment discontinuation.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib
Number analyzed (Participants) | 3014
Months | 13.5 [12.6 to 13.9]

5. Secondary Outcome: Response Rate (RR)
Description: RR was defined as the number (%) of participants with a best response (by Investigator assessment) of 'responding', regardless of the method of evaluation, and was based on a subset of the full analysis set consisting of subjects with at least one documented response assessment. RR was summarised together with the 95% CI.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 2900
Percentage of participants | 57.3 [55.5 to 59.2]

ADVERSE EVENTS:
Time Frame: From screening to progression follow-up [every 6 weeks +/- 1 week] relative to the date of enrolment until the end of study [up to 43 months]
Description: Safety of AZD9291 by assessment of SAEs, AEs of special interest (AESI) [Interstitial Lung Disease/pneumonitis-like events, and QTc prolongation events].
  This study did not collect all AEs; only SAEs, adverse events leading to dose modification, adverse events leading to treatment discontinuation and AESI were collected. Therefore non-serious AEs which did not lead to dose modification/discontinuation and were not AESIs are excluded from this table.
Arm/Group | Osimertinib
All-Cause Mortality (participants affected / at risk) | 1361/3014
Serious Adverse Events (participants affected / at risk) | 657/3014
Other Adverse Events (participants affected / at risk) | 380/3014
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib (N=3014)
Anaemia (Blood and lymphatic system disorders) | 4
Myelosuppression (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1
Blood disorder (Blood and lymphatic system disorders) | 1
Bone marrow disorder (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 9
Cardiac arrest (Cardiac disorders) | 6
Myocardial infarction (Cardiac disorders) | 4
Cardiac failure congestive (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 2
Cardiomyopathy (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Cardiac dysfunction (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Cardiotoxicity (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Hypertensive heart disease (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 4
Middle ear inflammation (Ear and labyrinth disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Cataract (Eye disorders) | 3
Dacryostenosis acquired (Eye disorders) | 2
Glaucoma (Eye disorders) | 2
Vomiting (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 4
Enteritis (Gastrointestinal disorders) | 4
Ascites (Gastrointestinal disorders) | 3
Chronic gastritis (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 3
Intestinal obstruction (Gastrointestinal disorders) | 3
Pancreatitis acute (Gastrointestinal disorders) | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Gingival ulceration (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Ischaemic enteritis (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Death (General disorders) | 34
Pyrexia (General disorders) | 12
Asthenia (General disorders) | 4
Sudden death (General disorders) | 4
Malaise (General disorders) | 3
Gait disturbance (General disorders) | 2
Multiple organ dysfunction syndrome (General disorders) | 2
Chest discomfort (General disorders) | 1
Condition aggravated (General disorders) | 1
Cyst (General disorders) | 1
Fatigue (General disorders) | 1
Granuloma (General disorders) | 1
Sudden cardiac death (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 5
Drug-induced liver injury (Hepatobiliary disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 3
Biliary colic (Hepatobiliary disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Liver injury (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 74
Upper respiratory tract infection (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 10
Respiratory tract infection (Infections and infestations) | 7
Bronchitis (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 6
Herpes zoster (Infections and infestations) | 5
Cellulitis (Infections and infestations) | 3
Osteomyelitis (Infections and infestations) | 3
Urosepsis (Infections and infestations) | 3
Device related infection (Infections and infestations) | 2
Empyema (Infections and infestations) | 2
Pulmonary sepsis (Infections and infestations) | 2
Abdominal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Complicated appendicitis (Infections and infestations) | 1
Diarrhoea infectious (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Enterobacter pneumonia (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Haemorrhagic fever (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Infective spondylitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Labyrinthitis (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 1
Nasal abscess (Infections and infestations) | 1
Otitis media acute (Infections and infestations) | 1
Peripheral nerve infection (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Respiratory tract infection bacterial (Infections and infestations) | 1
Scrub typhus (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 5
Femur fracture (Injury, poisoning and procedural complications) | 8
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 3
Spinal fracture (Injury, poisoning and procedural complications) | 3
Traumatic fracture (Injury, poisoning and procedural complications) | 3
Head injury (Injury, poisoning and procedural complications) | 2
Hip fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2
Multiple injuries (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Brain herniation (Injury, poisoning and procedural complications) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Electrocardiogram QT prolonged (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
Amylase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1
Influenza A virus test (Investigations) | 1
Lipase increased (Investigations) | 1
Troponin increased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 8
Decreased appetite (Metabolism and nutrition disorders) | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Malnutrition (Metabolism and nutrition disorders) | 3
Cachexia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7
Pathological fracture (Musculoskeletal and connective tissue disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Fracture pain (Musculoskeletal and connective tissue disorders) | 1
Malignant psoas syndrome (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 22
Headache (Nervous system disorders) | 6
Cerebral haemorrhage (Nervous system disorders) | 5
Transient ischaemic attack (Nervous system disorders) | 5
Cerebrovascular accident (Nervous system disorders) | 4
Epilepsy (Nervous system disorders) | 4
Cognitive disorder (Nervous system disorders) | 3
Lacunar infarction (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 2
Haemorrhage intracranial (Nervous system disorders) | 2
Haemorrhagic stroke (Nervous system disorders) | 2
Apraxia (Nervous system disorders) | 1
Basal ganglia infarction (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebellar ischaemia (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Facial paralysis (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Psychomotor skills impaired (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Thrombotic stroke (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Vascular headache (Nervous system disorders) | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Device dislocation (Product Issues) | 1
Completed suicide (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Breath holding (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Renal failure (Renal and urinary disorders) | 4
Haematuria (Renal and urinary disorders) | 3
Hydronephrosis (Renal and urinary disorders) | 2
Calculus urinary (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Renal injury (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Prostatic obstruction (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 49
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 9
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 17
Embolism (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 2
Venous thrombosis limb (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Superior vena cava occlusion (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib (N=3014)
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Neutropenia (Blood and lymphatic system disorders) | 16
Myelosuppression (Blood and lymphatic system disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 3
Pancytopenia (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 2
Ventricular extrasystoles (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Extrasystoles (Cardiac disorders) | 1
Nodal rhythm (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Blepharitis (Eye disorders) | 2
Cataract (Eye disorders) | 2
Ulcerative keratitis (Eye disorders) | 2
Conjunctival haemorrhage (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Swelling of eyelid (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Vitreoretinal traction syndrome (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 30
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 10
Stomatitis (Gastrointestinal disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Anal inflammation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 8
Pyrexia (General disorders) | 7
Fatigue (General disorders) | 4
General physical health deterioration (General disorders) | 4
Inflammation (General disorders) | 1
Influenza like illness (General disorders) | 1
Malaise (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Peripheral swelling (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 3
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Liver injury (Hepatobiliary disorders) | 1
Paronychia (Infections and infestations) | 11
Influenza (Infections and infestations) | 7
Herpes zoster (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 5
Atypical pneumonia (Infections and infestations) | 2
Cystitis (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 2
Herpes ophthalmic (Infections and infestations) | 2
Pneumonia viral (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2
Chemical burns of eye (Injury, poisoning and procedural complications) | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1
Electrocardiogram QT prolonged (Investigations) | 88
Platelet count decreased (Investigations) | 17
Aspartate aminotransferase increased (Investigations) | 10
Blood creatinine increased (Investigations) | 10
Alanine aminotransferase increased (Investigations) | 9
Neutrophil count decreased (Investigations) | 9
White blood cell count decreased (Investigations) | 8
Amylase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 2
Weight decreased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood pressure systolic increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Lipase increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 3
Abnormal loss of weight (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 3
Presyncope (Nervous system disorders) | 2
Balance disorder (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Demyelination (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Psychomotor skills impaired (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Azotaemia (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Nephropathy toxic (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Testicular cyst (Reproductive system and breast disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 10
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6
Skin toxicity (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Participants alive at the time of national reimbursement or site closure were no longer followed for survival and therefore prematurely censored for the OS, PFS, and TTD analysis, leading to less mature data. As the timing of reimbursement and study closure differed between countries, duration of follow-up between sites and countries differed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT02474355/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT02474355/SAP_001.pdf